CLINICAL TRIAL: NCT00267462
Title: Retrospective Review of Hypertrophic Myopathy in Children
Brief Title: Hypertrophic Myopathy in Children
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-034
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; hypertrophic Myopathy
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to identify the patients seen in our practice who are seen with Hypertrophic Myopathy diagnosis in order to better understand the presenting characteristics of their disease, the diagnostic testing to determine the diagnosis, the methods used to follow the disease progression and management practices used in caring for these patients. The objectives of this data review will be an analysis to determine if there is a methodology that will foster improved diagnostic speed and accuracy, and determine the best management practices based on outcomes in these patients.

DETAILED DESCRIPTION:
The charts of children followed at Sibley Heart Center of Children's Healthcare of Atlanta will be identified using the Mysis system and screening for the appropriate ICD-9 codes for the types of Hypertrophic Myopathy. These codes include: 425.1, 425.4, 425.7, 425.8, and 425.9. Screening will also be done for known anomalies that are associated with hypertrophic myopathy as seen in some syndromes and metabolic disorders.

Data Collection:

Age at presentation (DOB) History - Prenatal, Family, Current Surgical Procedures Physical Exam results EKG interpretation CXR results Echocardiography results MRI Results Holter monitors results Exercise testing results Radionuclear study results Spiral CT Study results Genetics Testing results Medication usage Enzyme replacement therapy usage Diagnostic laboratory results

Statistics:

A generalized linear model will be performed. Significance will be defined at P≤ 0.05.

Interim monitoring of accumulated data will be performed. One interim analysis will be performed after 3 months of accrual with additional analyses being performed at the end of data collection.

Demographic data will be summarized for all subjects. For each patient summary statistics will include the mean, standard deviation, frequency distribution, minimum, maximum and range.

ELIGIBILITY:
Inclusion Criteria:

* seen at Sibley Heart Center, Children's Healthcare of Atlanta
* diagnosed with Hypertrophic Myopathy

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Dooley, MD, Principal Investigator — Sibley Heart Center Cardiology at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States